CLINICAL TRIAL: NCT05489679
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Preliminary Anti-Tumor Activity of AC682 In Chinese Patients With ER+/HER2- Locally Advanced or Metastatic Breast Cancer
Brief Title: A Study of AC682 In Chinese Patients With ER+/HER2- Locally Advanced or Metastatic Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Voluntarily terminate the study since the sponsor's development strategy was adjusted.
Sponsor: Accutar Biotechnology Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AC682-002
Record Dates: First submitted 2022-07-15; First posted 2022-08-05 (Actual); Last update posted 2024-01-25 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer
Keywords: Estrogen receptor positive; ER positive; ER+; Human epidermal growth factor receptor 2 negative; HER2 negative; AC682; Phase I
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- AC682 (Experimental): This arm will evaluate AC682 monotherapy administered in 28-day cycles. The participants will participate in this dose escalation arm.
  Interventions: Drug: AC682

INTERVENTIONS:
Drug: AC682 — Participants will receive AC682 by mouth daily in 28-day cycles.

SUMMARY:
This clinical trial is evaluating AC682 in participants with estrogen receptor positive/human epidermal growth factor 2 negative (ER+/HER2-) locally advanced or metastatic breast cancer. The main goals of this study are to:

1. To evaluate the safety and tolerability of AC682
2. To evaluate the pharmacokinetic of AC682
3. To evaluate the preliminary anti-tumor activity of AC682

DETAILED DESCRIPTION:
This is a Phase I, open-label dose-escalation study of AC682, an orally available estrogen receptor degrader, given as a single agent.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be ≥18 years-of-age at the time of signing of the ICF
2. Histologically and/or cytologically confirmed advanced estrogen receptor positive (ER+) human epidermal growth factor 2 negative (HER2-) breast cancer
3. Female patients must be postmenopausal
4. At least 1 measurable lesion according to Response Evaluation Criteria in Solid Tumors (RECIST) Version 1.1 or at least 1 predominantly lytic bone lesion in the absence of measurable disease
5. Previously received at least 1 endocrine therapy regimen; concomitant use of cyclin-dependent kinase (CDK) 4/6 inhibitor(s) is acceptable; Previous chemotherapy is not required, but up to 2 prior regimens of cytotoxic chemotherapy is allowed.
6. Patients who have adequate organ functions at baseline

Exclusion Criteria:

1. Treatment with any of the following:

   systemic anti-cancer chemotherapy, biologic, or hormonal agent from a previous treatment regimen or clinical study within 4 weeks prior to the first dose of AC682; systemic small molecules from a previous treatment regimen or clinical study within 14 days or 5 half-lives (whichever is longer) prior to the first dose of AC682 (at least 10 days must have elapsed between the last dose of such agent and the first dose of study drug)
2. Received radiotherapy (including radioactive isotope therapy) within 4 weeks prior to the first dose of AC682
3. Major surgery (excluding placement of vascular access) within 4 weeks of first dose of AC682
4. With known metastasis to the brain
5. Any condition that impairs a patient's ability to swallow whole pills. Impairment of gastrointestinal function (GI) or GI disease or other condition at baseline that will interfere significantly with the absorption, distribution, or metabolism of AC682.
6. Use of prophylactic growth factors and blood transfusions ≤14 days prior to the first dose of AC682 and during dose limiting toxicity observation period

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2022-10-01 (Actual); Primary Completion 2023-09-28 (Actual); Study Completion 2023-09-28 (Actual)

PRIMARY OUTCOMES:
Incidence of dose limiting toxicities (DLTs) from AC682 monotherapy | 28 days
  Number of subjects with DLT
Incidence of treatment emergent adverse events(TEAEs) from AC682 monotherapy | Throughout the study completion, approximately 24 months
  Number of adverse events as characterized by type, frequency, seriousness, and relationship to AC682

SECONDARY OUTCOMES:
To determine the PK of AC682 after a single dose or multiple doses: | At predefined intervals throughout the study completion, approximately 24 months.
  Area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC(0-inf))
To determine the PK of AC682 after a single dose or multiple doses: | At predefined intervals throughout the study completion, approximately 24 months.
  Area under the concentration-time curve over the dosing interval (AUC(0-tau))
To determine the PK of AC682 after a single dose or multiple doses: | At predefined intervals throughout the study completion, approximately 24 months.
  Maximum plasma concentration (Cmax)
To determine the PK of AC682 after a single dose or multiple doses: | At predefined intervals throughout the study completion, approximately 24 months.
  Time to maximum plasma concentration (tmax)
To determine the PK of AC682 after a single dose or multiple doses: | At predefined intervals throughout the study completion, approximately 24 months.
  Terminal elimination half life (t1/2)
To evaluate the preliminary anti-tumor activity of AC682: | Throughout the study completion, approximately 24 months
  Objective Response Rate(ORR) using RECIST version 1.1
To evaluate the preliminary anti-tumor activity of AC682: | Throughout the study completion, approximately 24 months
  Clinical Benefit Rate (CBR) using RECIST version 1.1
To evaluate the preliminary anti-tumor activity of AC682: | Throughout the study completion, approximately 24 months
  Duration of Response (DoR) using RECIST version 1.1
To evaluate the preliminary anti-tumor activity of AC682: | Throughout the study completion, approximately 24 months
  Disease Control Rate (DCR) using RECIST version 1.1
To evaluate the preliminary anti-tumor activity of AC682: | Throughout the study completion, approximately 24 months
  Progression-free Survival (PFS) using RECIST version 1.1

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Site 1001, Beijing
  - Site 1003, Hangzhou
  - Site 1002, Tianjin